CLINICAL TRIAL: NCT01196676
Title: A Phase I, Randomized, Double- Blind, Placebo- Controlled, Single-center Study, to Assess the Safety, Tolerability and Pharmacokinetics of AZD4451 Following Single Ascending Oral Dose Administration in Healthy Subjects
Brief Title: Single Ascending Dose Study to Assess the Safety, Tolerability and Pharmacokinetics of AZD4451
Acronym: AZD4451 SAD
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Medical Science Director, AstraZeneca
Allocation: Randomized | Model: Single Group | Masking: Quadruple
Other Study IDs: D3600C00001
Record Dates: First submitted 2010-08-20; First posted 2010-09-08 (Estimated); Last update posted 2011-08-01 (Estimated); Status verified 2011-07

CONDITIONS: Bipolar Disorder
Keywords: AZD4451; Bipolar; depression
MeSH Terms: conditions — Bipolar Disorder; Depression

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): AZD4451
  Interventions: Drug: AZD4451
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD4451 — 1 mg capsules, 5 mg capsules, and 25 mg capsules
  Arms: 1
Drug: Placebo — 1 mg capsules, 5 mg capsules, and 25 mg capsules
  Arms: 2

SUMMARY:
This is a single ascending dose study to assess the safety, tolerability and pharmacokinetics of AZD4451.

ELIGIBILITY:
Inclusion Criteria:

* Provide a signed and dated, written informed consent prior to any study specific procedures being performed. including the genetic sampling and analyses. If a volunteer declines to participate in the genetic component of the study, there will be no penalty or loss of benefit to the volunteer. The volunteer will not be excluded from other aspects of the study described in this protocol.
* Healthy male and female (of non-childbearing potential) volunteers 18 to 55 years old inclusive with suitable veins for cannulation or repeated venipuncture.
* Females must have a negative pregnancy test at screening and on admission to the unit, must not be nursing and must be of non-childbearing potential, confirmed at screening by fulfilling one of the following criteria:
* Post-menopausal defined as amenorrhoea for at least 12 months following cessation of all exogenous hormonal treatments and with FSH levels in the laboratory defined post-menopausal range
* Documentation of irreversible surgical sterilization by hysterectomy, bilateral oophorectomy, or bilateral salpingectomy but not tubal ligation Male volunteers should be willing to use barrier contraception for example, condoms and spermicide, from the day of dosing until at least 3 months after dosing with the investigational product.
* Have a body mass index (BMI) between 19 and 30 kg/m2 (BMI <30.5 =30) and weigh at least 50 kg and no more than 100 kg inclusive.

Exclusion Criteria:

* History of gastrointestinal surgery (other than cholecystectomy or appendectomy) or unintentional rapid weight loss.
* A positive result on screening for serum hepatitis B surface antigen, hepatitis C antibody and human immunodeficiency virus (HIV).
* History of any of the following as judged by the Investigator: History of psychiatric disorders as defined in the Diagnostic and Statistical Manual of Mental Disorders text revision; Medically diagnosed depression in the 6 months prior to dosing; Bipolar disorder; Use of psychoactive medication (including mood stabilizers) in the 6 months prior to dosing; Electroconvulsive therapy in the 6 months prior to dosing; History of seizures 1 year prior to dosing; History of severe dystonic reaction to other drugs.
* History of syncope, fainting or of vasovagal reactions; history of arrhythmias, and/or postural hypotension. The inclusion of volunteers meeting the above criteria may be decided on a case-by-case basis after consultation between the Investigator and AZ CPA physician.
* History or presence of gastrointestinal, hepatic or renal disease or any other condition known to interfere with absorption, distribution, metabolism or excretion of drugs.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 63 (Estimated)
Dates: Start 2010-08; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
To assess the safety and tolerability of single ascending oral doses of AZD4451 by assessing AEs, vital signs, physical examinations, neurological examinations clinical laboratory parameters, Columbia Suicide Severity Rating Scale(CSSRS), EEGs and ECGs | Screening to end of study.

SECONDARY OUTCOMES:
To assess the pharmacokinetics of single ascending oral doses of AZD4451 by maximum plasma concentration (Cmax). | Predose, 30 min, 1 hr, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, 18, 24, 30, 48, and 72 hours postdose.
To evaluate and characterize the PK of AZD4451 and its metabolites AZ13263197 and AZ13263195 when given orally in single ascending doses by assessment of drug concentration in urine. | Urine will be collectioned for 72 hours post-dose. Pre-dose to 12 hours, 12-24, 24- 48 and 48-72 hours post-dose.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Smith, Study Director — AstraZeneca, LP, 1800 Concord Pike, Wilmington, DE; Ralph Schutz, Principal Investigator — Quintiles Phase I Services, 6700 West 115th Street, Overland Park, Kansas 66211
Locations (1):
- Research Site, Overland Park, Kansas, United States